CLINICAL TRIAL: NCT04412018
Title: An Investigation on the Effects of Icosapent Ethyl (VascepaTM) on Inflammatory Biomarkers in Individuals With COVID-19 (VASCEPA-COVID-19)
Brief Title: An Investigation on the Effects of Icosapent Ethyl (VascepaTM) on Inflammatory Biomarkers in Individuals With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Medical and Surgical Knowledge Translation Research Group (Other)
Collaborators: Amarin Corporation (Unknown); HLS Therapeutics, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00043601
Record Dates: First submitted 2020-05-29; First posted 2020-06-02 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: COVID-19; Inflammatory Response
MeSH Terms: conditions — COVID-19 | interventions — eicosapentaenoic acid ethyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Usual Care (No Intervention): Participants in this arm will continue with usual care
- Icosapent Ethyl (Experimental): Participants in this arm will take icosapent ethyl (4 g BID for 3 days, then 2 g BID for the subsequent 11 days)
  Interventions: Drug: Icosapent ethyl

INTERVENTIONS:
Drug: Icosapent ethyl — Icosapent ethyl (4 g BID for 3 days, then 2 g BID for the subsequent 11 days)
  Other Names: Vascepa
  Arms: Icosapent Ethyl

SUMMARY:
This is a 14-day long prospective, multi-site, two-armed, randomized, open-label study that will enroll approximately 100 adult outpatients in Canada who have received a positive SARS-CoV-2 test result within the preceding 72 hours. Participants will be randomized (1:1) to receive either icosapent ethyl (4 g BID for 3 days, then 2 g BID for the subsequent 11 days) or usual care. Blood samples will be collected to determine if icosapent ethyl use lowers circulating pro-inflammatory biomarkers.

ELIGIBILITY:
Inclusion Criteria:

1. Positive local SARS-CoV-2 test result within the preceding 72 hours
2. At least one of the following symptoms

   1. Fever
   2. Cough
   3. Sore throat
   4. Shortness of breath
   5. Myalgia

Exclusion Criteria:

1. Individuals currently participating in another interventional trial that will or may interfere with the primary outcome
2. Hospitalized individuals
3. Individuals who have a current medical condition for which life expectancy is less than 3 months
4. Individuals with a history of acute end-organ injury (e.g. myocardial infarction, stroke, hospitalization for acute lung, liver or kidney disease) within the last month
5. Individuals with active severe liver disease
6. Individuals with a history of acute or chronic pancreatitis
7. Women who are pregnant, may be pregnant, are planning on becoming pregnant, or are lactating
8. Women of child-bearing potential who are not using at least one form of highly effective (hormonal contraceptives [e.g. combined oral contraceptives, patch, vaginal ring, injectables, and implants]; intrauterine device or intrauterine system; tubal ligation or whose partner has had a vasectomy) and one effective (barrier methods such male condom, female condom, cervical cap, diaphragm, or contraceptive sponge) method of contraception
9. Individuals with a history of hemodynamic instability within past 72 hours including a systolic blood pressure of <95 mmHg and/or a diastolic blood pressure of <50 mmHg
10. Individuals with known hypersensitivity to fish and/or shellfish, or ingredients of IPE
11. Individuals with any other condition which, in the opinion of the Investigator, would place the participant at increased risk, preclude obtaining voluntary consent or confound the objectives of study
12. Individuals who are unable to swallow IPE capsules whole

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2020-11-06 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Change in hs-CRP levels from the randomization visit (Day 1) to the Day 14 visit | 14 days

SECONDARY OUTCOMES:
Change in D-dimer levels from the randomization visit (Day 1) to the Day 14 visit | 14 days
Change in erythrocyte sedimentation rate from the randomization visit (Day 1) to the Day 14 visit | 14 days
Change in complete blood count from the randomization visit (Day 1) to the Day 14 visit | 14 days
Change in differential count from the randomization visit (Day 1) to the Day 14 visit | 14 days
Change in serum albumin levels from the randomization visit (Day 1) to the Day 14 visit | 14 days
Change in neutrophil-to-lymphocyte ratio (NLR) from the randomization visit (Day 1) to the Day 14 visit | 14 days
Change in systemic immune-inflammation index from the randomization visit (Day 1) to the Day 14 visit | 14 days

OTHER OUTCOMES:
Change in FLU-PRO scores from the screening visit to the Day 14 visit | 14 days
  Response options will be along one of the following formats:
  (i) 5-point Likert scale with answers ranging from (a) "Not at all" to "Very much" and (b) "Never" to "Always" (ii) Quantitative with answers ranging from "0 times" or "4 or more times" (iii) Binary response format (Yes or No)
World Health Organization Symptom Severity Scale | 14 days
  Response options will range from 0 to 6 with a higher value indicating a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Subodh Verma, MD, PhD, Principal Investigator — Canadian Medical and Surgical Knowledge Translation Research Group
Locations (1):
- North York Diagnostic and Cardiology Clinic, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kosmopoulos A, Bhatt DL, Meglis G, Verma R, Pan Y, Quan A, Teoh H, Verma M, Jiao L, Wang R, Juliano RA, Kajil M, Kosiborod MN, Bari B, Berih AA, Aguilar M, Escano A, Leung A, Coelho I, Hibino M, Diaz R, Mason RP, Steg PG, Simon T, Go AS, Ambrosy AP, Choi R, Kushner AM, Leiter LA, Al-Omran M, Verma S, Mazer CD. A randomized trial of icosapent ethyl in ambulatory patients with COVID-19. iScience. 2021 Sep 24;24(9):103040. doi: 10.1016/j.isci.2021.103040. Epub 2021 Aug 26. PMID 34462732